CLINICAL TRIAL: NCT02540629
Title: Implementation of Gold Standard EMS CPR Programs for 2% Improvement in Survival Rates of Out-of-Hospital Cardiac Arrest in a Metropolitan City
Acronym: 2% Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Human resource change in Research investigators and Seoul Fire Department
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Do Shin, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-EM-2015-3
Record Dates: First submitted 2015-08-06; First posted 2015-09-04 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Cardiopulmonary resuscitation; Emergency Medicine
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Before intervention (No Intervention): The before intervention group will include patients from January, 2013 through December, 2014, as to refer to the historic control population who did not receive any of study interventions.
- After intervention (Experimental): The main study phase was planned to begin in January, 2016 through December, 2017, for a total of two years. Patients during the main study phase will have received one or more study interventions as applicable. However, because we could not continue our project in 2017, we changed after period. We included implementation period (2015) in after period. Therefore, final after period begins in January 2015 to December 2016.
  Interventions: Procedure: Bundled EMS CPR approach including dispatcher-assisted CPR, 3-person team CPR, and feedback CPR monitoring device

INTERVENTIONS:
Procedure: Bundled EMS CPR approach including dispatcher-assisted CPR, 3-person team CPR, and feedback CPR monitoring device — Gold standard EMS CPR refers to our bundled approach to providing high quality EMS CPR through one or more intervention(s) as applicable including 1) dispatcher-assisted CPR, 2) multi-tiered team CPR, and 3) feedback CPR.
  Arms: After intervention

SUMMARY:
This study aims to improve the survival rate of out-of-hospital cardiac arrest patients by 2% through a bundle of three intervention measures including: 1) dispatcher-assisted CPR, 2) multi-tiered response team CPR, and 3) feedback CPR.

DETAILED DESCRIPTION:
The project aims to implement gold standard emergency medical services (EMS) cardiopulmonary resuscitation (CPR) programs, which will result in increased bystander CPR, reduced EMS response time, and high quality CPR during prehospital resuscitation through a bundled approach including 1) dispatcher-assisted CPR (DA-CPR), 2) multi-tiered response team CPR, and 3) feedback CPR.

The DA-CPR program aims to contribute to improved bystander CPR rate and reduced EMS response time interval through rigorous monitoring of cardiac arrest detection at primary call receiving stage as well as increased number of dispatcher-assisted CPR instruction initiation in the target time of 90 seconds. The Team CPR protocol will render synergetic efforts among participating EMS personnel from both basic life support (BLS) and advanced life support (ALS) units within the new tiered dispatch system and subsequently deliver uninterrupted CPR to out-of-hospital cardiac arrest (OHCA) patients before hospital arrival. The feedback CPR monitoring and quality assurance program will contribute to high quality CPR delivered to the patients on the scene as well as during transport.

ELIGIBILITY:
Inclusion Criteria:

* EMS-assessed OHCA
* Cardiac etiology
* Above 15 years of age

Exclusion Criteria:

* Patients who do not receive EMS resuscitation
* Patients with signs of evident death (decapitation, evident livor mortis or rigor mortis)
* Do-Not-Resuscitate cases
* Pregnant patients
* Patients whom the mechanical devices cannot be applied to

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12670 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional EMS CPR (2013-2014, 2 Years): Conventional EMS CPR group will include patients from January, 2013 through December, 2014, as to refer to the historic control population who did not receive any of study interventions.
- Bundled EMS CPR (2015-2016, 2 Years): The main study phase will begin in January, 2015 through December, 2016, for a total of two years. Patients during the main study phase will have received one or more study interventions as applicable.
  Bundled EMS CPR approach including dispatcher-assisted CPR, 3-person team CPR, and feedback CPR monitoring device: Gold standard EMS CPR refers to our bundled approach to providing high quality EMS CPR through one or more intervention(s) as applicable including 1) dispatcher-assisted CPR, 2) multi-tiered team CPR, and 3) feedback CPR.
Period: Overall Study
Arm/Group | Conventional EMS CPR (2013-2014, 2 Years) | Bundled EMS CPR (2015-2016, 2 Years)
Started | 6201 | 6469
Completed | 6201 | 6469
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional EMS CPR (2013-2014, 2 Years) | Bundled EMS CPR (2015-2016, 2 Years) | Total
Number analyzed (Participants) | 6201 | 6469 | 12670
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [58 to 80] | 73 [59 to 81] | 72 [59 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2227 | 2344 | 4571
  Male | 3974 | 4125 | 8099
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6201 | 6469 | 12670
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 6201 | 6469 | 12670
Public place [Count of Participants; unit: Participants] | 1180 | 1261 | 2441
Witnessed [Count of Participants; unit: Participants] | 3119 | 3353 | 6472
Bystander CPR [Count of Participants; unit: Participants]
  No bystander CPR | 2739 | 2526 | 5265
  Bystander CPR with dispatcher assistace | 2357 | 2866 | 5223
  Bystander CPR without dispatcher assistace | 1105 | 1077 | 2182
Initial shockable rhythm [Count of Participants; unit: Participants] | 696 | 719 | 1415
Multi-tier response [Count of Participants; unit: Participants]
  Single tier | 6201 | 4047 | 10248
  Multi-tier with ambulance | 0 | 2080 | 2080
  Multi-tier with fireengine | 0 | 342 | 342
Feedback CPR [Count of Participants; unit: Participants] — Using feed-back CPR device
  - CPR using equipment to measure CPR quality (depth and rate)
  Participants | 1628 | 3978 | 5606
Prehospital ROSC [Count of Participants; unit: Participants] — Number of participants with prehospital return of spontaneous circulation (ROSC before arriving hospital)
  Participants | 471 | 701 | 1172

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Survival to Hospital Discharge
Description: Number of EMS-assessed out-of-hospital cardiac arrest patients who survive to hospital discharge will be recorded.
Time Frame: At hospital discharge, up to 28 weeks from hospital admission
Measure: Count of Participants; unit: Participants
Groups:
- Conventional EMS CPR: Conventional EMS CPR group will include patients from January, 2013 through December, 2014, as to refer to the historic control population who did not receive any of study interventions.
- Bundled EMS CPR: The main study phase will begin in January, 2015 through December, 2016, for a total of two years. Patients during the main study phase will have received one or more study interventions as applicable.
  Bundled EMS CPR approach including dispatcher-assisted CPR, 3-person team CPR, and feedback CPR monitoring device: Gold standard EMS CPR refers to our bundled approach to providing high quality EMS CPR through one or more intervention(s) as applicable including 1) dispatcher-assisted CPR, 2) multi-tiered team CPR, and 3) feedback CPR.
Arm/Group | Conventional EMS CPR | Bundled EMS CPR
Number analyzed (Participants) | 6201 | 6469
Participants | 594 | 707
Statistical Analysis 1: Comparison: Conventional EMS CPR vs Bundled EMS CPR; Test type: Equivalence — Chi-squared test; p = 0.01, Chi-squared

2. Secondary Outcome: Number of Participants With Good Neurological Recovery at Discharge
Description: Number of EMS-assessed out-of-hospital cardiac arrest patients who survive to hospital discharge and has cerebral performance category 1 or 2 will be recorded.
Time Frame: At hospital discharge, up to 28 weeks from hospital admission
Measure: Count of Participants; unit: Participants
Groups:
- Bundled EMS CPR: The main study phase will begin in January, 2016 through December, 2017, for a total of two years. Patients during the main study phase will have received one or more study interventions as applicable.
  Bundled EMS CPR approach including dispatcher-assisted CPR, 3-person team CPR, and feedback CPR monitoring device: Gold standard EMS CPR refers to our bundled approach to providing high quality EMS CPR through one or more intervention(s) as applicable including 1) dispatcher-assisted CPR, 2) multi-tiered team CPR, and 3) feedback CPR.
Arm/Group | Conventional EMS CPR | Bundled EMS CPR
Number analyzed (Participants) | 6201 | 6469
Participants | 334 | 441

ADVERSE EVENTS:
Time Frame: At hospital discharge, up to 28 weeks from hospital admission
Arm/Group | Conventional EMS CPR | Bundled EMS CPR
All-Cause Mortality (participants affected / at risk) | 5607/6201 | 5762/6469
Serious Adverse Events (participants affected / at risk) | 0/6201 | 0/6469
Other Adverse Events (participants affected / at risk) | 0/6201 | 0/6469

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT02540629/Prot_SAP_000.pdf